CLINICAL TRIAL: NCT02340351
Title: Auricular Acupuncture Versus Progressive Muscle Relaxation in Patients With Anxiety Disorders or Major Depressive Disorder.
Brief Title: Auricular Acupuncture vs. Progressive Muscle Relaxation in Patients With Anxiety Disorders or Major Depressive Disorder.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKE-Psych-Aku-08-14
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Anxiety Disorders; Depressive Disorder, Major
Keywords: acupuncture; auricular acupuncture; NADA; anxiety; depression
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder, Major; Depression | interventions — Acupuncture, Ear; Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Auricular acupuncture (Active Comparator): Within this arm, patients were treated with auricular acupuncture according to the NADA protocol. Each setting involved not more than eight patients at a time and was performed in a sitting position. Each session lasted 30 minutes and took place twice a week over a period of 4 weeks.
  Interventions: Device: Auricular acupuncture
- Progressive muscle relaxation (Active Comparator): Within this arm, patients were treated with who chose treatment with progressive muscle relaxation. Each setting involved not more than eight patients at a time and was performed in a sitting position. Each session lasted 30 minutes, took place twice a week over a period of 4 weeks.
  Interventions: Procedure: Progressive muscle relaxation

INTERVENTIONS:
Device: Auricular acupuncture — Auricular acupuncture according to the the NADA protocol includes the needling of five specific acupuncture points on both ears: point 51 (= Sympathetic point), point 55 (= Shen Men), point 95 (= Kidney point), point 97 (= Liver point) and point 101 (= Lung point). All points were acupunctured with fine sterile single use steel needles with the size of 0.25 x 20 millimetres. The needles were inserted about 2-3 millimetres, so that the needle point pierces the skin and is just positioned in the cartilage of the ear. They remained in position for 30 minutes.
  Arms: Auricular acupuncture
Procedure: Progressive muscle relaxation — Progressive muscle relaxation was carried out by the method of Bernstein and Borkovec. All participants were asked to close eyes while sitting comfortably. Each group session included 16 main exercises of consciously tensing and relaxing specific groups of muscles.
  Arms: Progressive muscle relaxation

SUMMARY:
The purpose of this study is to determine whether auricular acupuncture (AA) according to the NADA protocol and progressive muscle relaxation (PMR) differ in their effectiveness of treating people with anxiety disorders or major depressive disorder. We hypothesized, that both treatments show significant effects in alleviating the examined items (tension, anxiety, anger/aggression and state ofr mood) and that there is no significant difference between these two treatments.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether auricular acupuncture according to the NADA protocol and progressive muscle relaxation differ in their effectiveness of treating people with anxiety disorders (AD) or major depressive disorder (MDD).

In this study, acupuncture was executed according to the NADA protocol: a standardized and comparable method of auricular acupuncture (AA) with ease of application and limited adverse reactions, which seems to have high acceptance among psychiatric patients. The NADA (National Acupuncture Detoxification Association) protocol includes the needling of five specific acupuncture points on both ears.

As a comparative relaxation treatment, progressive muscle relaxation (PMR) was applied in our study. It has been well established for many decades, especially for the treatment of severe states of physical and mental tension, which is a common symptom of anxiety disorders and depression. Many studies also suggest its potential utility in the treatment program of many other illnesses, which are associated with conditions of anxiety and depression, such as schizophrenia, sleeping disorders, endometriosis, atopic dermatitis or cancer.

The main aim of this study was to examine the effectiveness of AA according to the NADA protocol versus PMR in patients with AD or MDD. We hypothesized, that both treatments show significant effects in alleviating the examined items (tension, anxiety, anger/aggression and state ofr mood) and that there is no significant difference between these two treatments. In order to increase the patients´ treatment acceptance and compliance, this study was set up in an open design in which each patient was freely able to choose between both treatments.

ELIGIBILITY:
Inclusion Criteria:

* patient at our psychiatric ward or day-hospital
* meeting the DSM-IV diagnostic criteria for the primary diagnosis of an anxiety disorder oder major depressive disorder

Exclusion Criteria:

* ear infection
* anamnestic substance abuse or positive drug screening
* taking opioid analgesics
* suffering from schizophrenic or organic cerebral psychosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2007-07; Primary Completion 2009-03 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Mean VAS scores of anxiety, tension, anger/aggression and mood before and after treatment within each treatment group at week 1. | 1 week
  VAS are rated as follows: ´tension´, ´anxiety´, ´anger/aggression´: VAS 0 = none, 100 = most imaginable; ´mood´: VAS 0 = bad, 100 = good.
Mean VAS scores of anxiety, tension, anger/aggression and mood before and after treatment within each treatment group at week 2. | week 2
  VAS are rated as follows: ´tension´, ´anxiety´, ´anger/aggression´: VAS 0 = none, 100 = most imaginable; ´mood´: VAS 0 = bad, 100 = good.
Mean VAS scores of anxiety, tension, anger/aggression and mood before and after treatment within each treatment group at week 3. | week 3
  VAS are rated as follows: ´tension´, ´anxiety´, ´anger/aggression´: VAS 0 = none, 100 = most imaginable; ´mood´: VAS 0 = bad, 100 = good.
Mean VAS scores of anxiety, tension, anger/aggression and mood before and after treatment within each treatment group at week 4. | week 4
  VAS are rated as follows: ´tension´, ´anxiety´, ´anger/aggression´: VAS 0 = none, 100 = most imaginable; ´mood´: VAS 0 = bad, 100 = good.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Muhtz, MD, Principal Investigator — Department of Psychosomatic Medicine and Psychotherapy, University Medical Center Hamburg-Eppendorf & Schoen Klinik Hamburg-Eilbek, Hamburg, Germany